CLINICAL TRIAL: NCT04137484
Title: Evaluation of a Patient Blood Management Program in Total Hip or Total Knee Arthroplasty
Brief Title: Patient Blood Management Program in Total Hip or Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0484
Record Dates: First submitted 2019-10-14; First posted 2019-10-24 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Knee Arthropathy; Hip Arthropathy
Keywords: Patient Blood Management Program; Transfusion; Postoperative anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Total hip and knee arthroplasty are among the most common surgical procedures for which blood transfusion is prescribed. Patient blood management program has been proposed to decrease the need for transfusion. This program involve three pillars: preoperative improvement of erythropoiesis, intraoperative reduction of bleeding and postoperative management of anemia.

Among the different steps of this program, reduction of bleeding and optimization of anemia are gaining popularity, but preoperative improvement of erythropoiesis is underused. The preoperative step of the blood management program is not systematically used because it requires a complex organization, is considered expensive, and finally because the others available techniques to reduce blood transfusion are easier to implement.

The aim of this study was to assess, within a patient blood management program, the effectiveness of erythropoietin on reducing allogenic blood transfusion and anemia in patients requiring elective total hip or knee arthroplasty. "

DETAILED DESCRIPTION:
This is a post-hoc analysis using part of the patients involved in the Cross Iron Study (Anesthesiology. 2018 Oct;129(4):710-720 ) Included patients were all the patients scheduled for elective primary total hip or knee arthroplasty and assessed by an anesthesiologist involved in the Cross Iron Study. Exclusion criteria were pregnancy, age under 18 years old, systemic infection, bilateral arthroplasty, revision arthroplasty, and participation in a preoperative autologous donation program.

This was a observational study. The patient blood management program included: erythropoietin with iron supplementation if preoperative hemoglobin was lower than 13 g/dl; tranexamic acid during surgery; intravenous iron postoperatively and use of prespecified thresholds for homologous blood transfusion. Blood transfusion and anemia were assessed until day 5 or discharge, whichever came first. Major thromboembolic or cardiovascular events were assessed during admission and one month after discharge.

ELIGIBILITY:
Inclusion Criteria:

* patient from the flow chart of the Cross Iron Study (Anesthesiology. 2018 Oct;129(4):710-720 )
* patient scheduled for elective primary total hip or knee arthroplasty

Exclusion criteria:

* pregnancy patient,
* patient under 18 years old
* systemic infection
* bilateral arthroplasty
* revision arthroplasty,
* participation in a preoperative autologous donation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the flow chart of the Cross Iron Study (Anesthesiology. 2018 Oct;129(4):710-720 ) Included patients were all the patients scheduled for elective primary total hip or knee arthroplasty and assessed by an anesthesiologist involved in the Cross Iron Study.
Sampling Method: Non-Probability Sample
Enrollment: 723 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Blood transfusion induced by postoperative anemia at hospital discharge | before the anesthesia consultation, the day before surgery, and after surgery at day 1, day 3 and day 5 if still admitted
  Hemoglobin was systematically assessed during surgery and after surgery at day 1, day 3 and day 5 if still admitted. The Hb thresholds for homologous blood transfusion used during the intra- and postoperative period were 7 g/dl in healthy patients in the absence of physical activity, 8 to 9 g/dl in the presence of physical activity (early rehabilitation) or in patients with cardiovascular disease, and 10 g/dl in patients with cardiac or coronary insufficiency.
Blood transfusion induced by postoperative anemia at hospital discharge | before the anesthesia consultation, the day before surgery, and after surgery at day 1, day3 and day 5 if still admitted
  Hemoglobin was systematically assessed during surgery and after surgery at day 1, day 3 and day 5 if still admitted. The Hb thresholds for homologous blood transfusion used during the intra- and postoperative period were 7 g/dl in healthy patients in the absence of physical activity, 8 to 9 g/dl in the presence of physical activity (early rehabilitation) or in patients with cardiovascular disease, and 10 g/dl in patients with cardiac or coronary insufficiency.

SECONDARY OUTCOMES:
Rate of major complications one month after surgery | admission in intensive care unit, and death were reported on day 3, on day 5 if still admitted, and one month after surgery at the routine postoperative surgical consultation
  Major complications including thromboembolic events, cardiac or respiratory failure, admission in intensive care unit, and death were reported on day 3, on day 5 if still admitted, and one month after surgery at the routine postoperative surgical consultation

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BIBOULET, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC